CLINICAL TRIAL: NCT01189682
Title: Impact of Tegaderm HP and Tegaderm CHG in Major Catheter Related Infections and Dressing Detachment in ICU Patients a Prospective Randomized Study
Brief Title: Impact of Tegaderm HP and CHG in Major Catheter Related Infections and Dressing Detachment
Acronym: DRESSING2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-A01184-53
Record Dates: First submitted 2010-05-25; First posted 2010-08-27 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2012-09

CONDITIONS: Catheter-Related Infections
Keywords: catheter; dressing; chlorhexidine; Patient admitted in ICU with a CVC or art. catheter
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tegaderm HP (Active Comparator)
  Interventions: Procedure: Tegaderm, Tegaderm HP, Tegaderm CHG
- Tegaderm (Placebo Comparator)
  Interventions: Procedure: Tegaderm, Tegaderm HP, Tegaderm CHG
- Tegaderm CHG (Active Comparator)
  Interventions: Procedure: Tegaderm, Tegaderm HP, Tegaderm CHG

INTERVENTIONS:
Procedure: Tegaderm, Tegaderm HP, Tegaderm CHG — dressings on catheters
  Other Names: Tegaderm; Tegaderm HP; tegaderm CHG

SUMMARY:
Catheter related infection is a frequent and life threatening event in ICU. A chlorhexidine impregnated sponge has been proven to reduce the rate of major catheter related infections in ICU patients (HR=0.39, p=0.03) (Timsit Jama 2009). However, dressings are detached in 40% of cases before planned changes and the rate of unplanned dressing is significantly associated with the major catheter related infections.

Primary objective: To demonstrate that Tegaderm CHG, a new CHG impregnated dressing decrease the rate of major catheter related infection as compared to non impregnated dressings and to demonstrate that highly adhesive dressing decrease the rate of detached dressings.

Secondary objectives:

* To demonstrate that the use of high performance dressing decrease the rate of unstuck dressing and the rate of catheter infections.
* To evaluate the tolerance of CHG impregnated gel dressings (Tegaderm CHG).
* To calculate the cost saving of each dressings

DETAILED DESCRIPTION:
Inclusion criteria: Patients older than 18 years old with central venous who need a central vein and/or an arterial catheter for an expected duration of more than 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old with a central venous catheter or arterial catheter installed in the study departement for a maximum for 24 hours

Exclusion Criteria:

* pulmonary arterial catheter
* antiseptic-impregnated catheter
* hemodialysis catheter
* chlorhexidine allergy
* emergency catheter without surgical asepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Risk of major catheter infection between Group 1 and Group 2+3 assessed by an independent blind expert panel | 48 hours after catheter removal or ICU discharge (10 days on average)
  The patients were followed 48h after catheter removal or discharge. Average follow up of 10 days.

SECONDARY OUTCOMES:
dressing detachment : rate of unplanned dressing between Tegaderm CHG, Tegaderm HP and Tegaderm | until catheter removal or ICU discharge (8 days on average)
Comparison of Group 1 to group 2+3 : catheter colonization, CR-BSI, cutaneous colonization at catheter removal, cost | 48 hours after catheter removal or ICU discharge (10 days on average)

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT Jean-François, PU/PH, Principal Investigator — Unit Intensive care
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Valette X, Daubin C, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable model predicting the required catheter dwell time among mechanically ventilated critically ill patients in three randomized trials. Ann Intensive Care. 2023 Jan 16;13(1):5. doi: 10.1186/s13613-023-01099-9. PMID 36645531
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Ruckly S, Souweine B, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable prediction model of central venous catheter-tip colonization in a cohort of five randomized trials. Crit Care. 2022 Jul 7;26(1):205. doi: 10.1186/s13054-022-04078-x. PMID 35799302
- [Derived] Buetti N, Ruckly S, Schwebel C, Mimoz O, Souweine B, Lucet JC, Timsit JF. Chlorhexidine-impregnated sponge versus chlorhexidine gel dressing for short-term intravascular catheters: which one is better? Crit Care. 2020 Jul 23;24(1):458. doi: 10.1186/s13054-020-03174-0. PMID 32703235
- [Derived] Buetti N, Ruckly S, Lucet JC, Bouadma L, Schwebel C, Mimoz O, Timsit JF. Ultrasound guidance and risk for intravascular catheter-related infections among peripheral arterial catheters: a post-hoc analysis of two large randomized-controlled trials. Ann Intensive Care. 2020 Jul 8;10(1):89. doi: 10.1186/s13613-020-00705-4. PMID 32643100
- [Derived] Maunoury F, Motrunich A, Palka-Santini M, Bernatchez SF, Ruckly S, Timsit JF. Cost-Effectiveness Analysis of a Transparent Antimicrobial Dressing for Managing Central Venous and Arterial Catheters in Intensive Care Units. PLoS One. 2015 Jun 18;10(6):e0130439. doi: 10.1371/journal.pone.0130439. eCollection 2015. PMID 26086783
- [Derived] Timsit JF, Bouadma L, Mimoz O, Parienti JJ, Garrouste-Orgeas M, Alfandari S, Plantefeve G, Bronchard R, Troche G, Gauzit R, Antona M, Canet E, Bohe J, Herrault MC, Schwebel C, Ruckly S, Souweine B, Lucet JC. Jugular versus femoral short-term catheterization and risk of infection in intensive care unit patients. Causal analysis of two randomized trials. Am J Respir Crit Care Med. 2013 Nov 15;188(10):1232-9. doi: 10.1164/rccm.201303-0460OC. PMID 24127770
- [Derived] Timsit JF, Mimoz O, Mourvillier B, Souweine B, Garrouste-Orgeas M, Alfandari S, Plantefeve G, Bronchard R, Troche G, Gauzit R, Antona M, Canet E, Bohe J, Lepape A, Vesin A, Arrault X, Schwebel C, Adrie C, Zahar JR, Ruckly S, Tournegros C, Lucet JC. Randomized controlled trial of chlorhexidine dressing and highly adhesive dressing for preventing catheter-related infections in critically ill adults. Am J Respir Crit Care Med. 2012 Dec 15;186(12):1272-8. doi: 10.1164/rccm.201206-1038OC. Epub 2012 Oct 4. PMID 23043083